CLINICAL TRIAL: NCT04776226
Title: Impact of Pots-stroke Depression Treatment on Stroke Recurrence
Brief Title: Post-stroke Depression Treatment Effect on Stroke Recurrence
Acronym: STROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Emre Kumral, Prof. Dr. MD, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EU-2018/55
Record Dates: First submitted 2021-01-24; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Stroke Recurrence; Cardiovascular Events; Depression
Keywords: Depression; Treatment; Stroke; Myocardial infarction
MeSH Terms: conditions — Depression; Stroke; Myocardial Infarction | interventions — Citalopram

STUDY DESIGN:
Intervention Model Description: Three-site, prospective, nonrandomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: There is no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients without depression (No Intervention): This group included patients without depression during enrollment of the cases.
- Depressive patients with treatment (Experimental): This group included patients wit depression but with treatment during enrollment of the cases.
  Interventions: Drug: Citalopram
- Depressive patients wihout treatment (No Intervention): This group included patients without depression but withou treatment during enrollment of the cases.

INTERVENTIONS:
Drug: Citalopram — Antidepressant use in patients with depression
  Other Names: Treatment group; Nontreatment group
  Arms: Depressive patients with treatment

SUMMARY:
It is not clear whether depresssion can predispose, or precipitate stroke recurrence in patients with stroke. We sought the relationship of post stroke depression with stroke recurrence.

DETAILED DESCRIPTION:
A large body of evidence suggests that depression is associated with a increased risk of many chronic diseases, including hypertension, diabetes, stroke and particularly coronary heart disease. Post stroke depression (PSD) may develop as a result of vascular disease. A previous meta-analysis showed that depression significantly increased the risk of development of stroke, and this increase was probably independent of other risk factors, including hypertension and diabetes.

Clarifying this issue has important implications; if depression increases the risk of development of recurrent stroke, so treating PSD might decrease the occurrence of recurrent stroke. To our knowledge there is no study attempting to clarify the relationship between PSD treatment and stroke recurrence. To fill these gap, we systematically conducted a study to assess whether PSD is associated with recurrent stroke, cardiovascular events or death. Thus, in the current study, three different arms of follow-up of patients with first-ever stroke, were used to predict the outcome over 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

• Patients who met DSM-IV and V criteria for depression

Exclusion Criteria:

* Severe or unstable medical disorders (eg, myocardial infarction within past 3 months, end-stage cancer, decompensated cardiac failure)
* Known primary neurological disorders including dementia, delirium, Parkinson disease, brain tumors, multiple sclerosis, seizure disorder
* Drugs (eg, systemic steroids)
* Pancreatic cancer, uncorrected hypothyroidism
* Current suicidal risk
* Use of psychotropic prescription or nonprescription drugs, certain hypnotics
* Mini-Mental State Examination (MMSE) score of 21 or lower

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1230 (Actual)
Dates: Start 2017-02-11 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Stroke recurrence | 12 months
  Standard World Health Organization definitions were used for recurrent stroke

SECONDARY OUTCOMES:
Cardiovascular Event | 12 months
  Cardiovascular events were defined and recorded over the study period if they had at least one of the following: myocardial infarction; unstable angina; angina; percutaneous coronary intervention; or coronary artery bypass graft surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Nezih Özdemir, MD, Principal Investigator — Ege University Scool of Medicine
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
* Individual deidentified participant data are available, including data dictionaries. .Data were entered into the registry between April 2018 and December 2019.
  * Other documents are available (e.g., study protocol, statistical analysis plan).
Supporting Information: Study Protocol, SAP
Time Frame: 12 months
Access Criteria: The data will be shared with anyone on reasonable reason.